CLINICAL TRIAL: NCT03929315
Title: A Prospective Randomised Control Trial of Competency Metrics and Educational Interventions in the Learning of One Lung Ventilation Techniques in Children Using Low-cost 3D Printed Tracheo-bronchial Models Among Pediatric Anesthesia Trainees
Brief Title: 3D OLV Training Intervention for Pediatric Anesthesia Trainees
Status: Withdrawn | Type: Observational
Why Stopped: COVID made it difficult to access the materials and participants required for this study
Sponsor: Clyde Matava (Other)
Responsible Party: Sponsor-Investigator, Clyde Matava, Anesthesiologist, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Other Study IDs: 1000057104
Record Dates: First submitted 2019-04-15; First posted 2019-04-26 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia
Keywords: one lung ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-spaced learning: Learning/testing sessions will take place within 30 minutes of one another
  Interventions: Behavioral: OLV technique on tracheo-bronchial model
- Spaced learning: Learning/testing sessions will take place 1 week after one another
  Interventions: Behavioral: OLV technique on tracheo-bronchial model

INTERVENTIONS:
Behavioral: OLV technique on tracheo-bronchial model — Models will range in size from 6 yrs to 6 weeks.

SUMMARY:
One lung ventilation (OLV) in neonates and children is an advanced skill that is necessary for delivery of safe and quality anesthetic care. The current model of training for OLV in the paediatric patient is composed of the apprenticeship model. Trainees learn the techniques of doing the procedure when they encounter a case that allows for it. The model of training is often inadequate for mastery of skills such as OLV as children in this population often have severe debilitating disease often requiring the most experienced anesthesiologist to perform OLV. This limits the training exposure of anesthesia trainees.

DETAILED DESCRIPTION:
Each participant will be subjected to three learning sessions on a 6 year old tracheo-bronchial model. Learning will either be spaced (1 week between learning/testing sessions) or non-spaced (30 minutes between learning/testing sessions). They will have 20 minutes to practice on this model before they are asked to perform the OLV on a younger tracheo-bronchial model (2 yrs, 3 months, 6 weeks). After each testing session, the participants will be provided with feedback. After all learning/testing sessions take place, the participants will be asked to complete a retention test on the 6 week old model six weeks after their last session.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric residents and fellows from the Hospital for Sick Children, Toronto

Exclusion Criteria:

* Refusal to participate in study
* Previous experience with at most two OLV in children
* Previous experience with at most two OLV in manikins

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pediatric anesthesia trainees at the Hospital for Sick Children, Toronto
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Time | Day 1, after each learning session
  Seconds it took for correct placement of OLV
Time | Week 6 or 9
  Seconds in took for correct placement of OLV

SECONDARY OUTCOMES:
Attempts | Week 6 or 9
  Number of attempts per procedure
Wrong entry | Week 6 or 9
  Number of entries into wrong bronchus
Red-outs | Week 6 or 9
  Number of red-outs
Wall collisions | Week 6 or 9
  Number of wall collisions
Qualitative endoscopic assessment | Week 6 or 9
  Measured using Global Rating Scale of Fibreoptic Bronchoscope Manipulation, on a scale of 4-20, where 4=novice and 20=expert
Overall rating of performance | Week 6 or 9
  Measured using Visual Analogue Scale, on a scale of 0-100 where 0=novice and 100=expert
Satisfaction with task load | Day 1 or Weeks 1-3
  Measured using Task Load Index, on a scale of 0-100, where 0=very low and 100=very high
Satisfaction with usability | Day 1 or Weeks 1-3
  Measured using System Usability Scale, on a scale of 5-50

CONTACTS AND LOCATIONS:
Overall Officials: Clyde Matava, Principal Investigator — Anesthesiologist-in-Cheif
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No